CLINICAL TRIAL: NCT00678106
Title: A Phase 1, Open Label, Single Dose Study To Investigate The Pharmacokinetics, Safety And Tolerability Of Dalbavancin In Hospitalized Adolescents, Aged 12 Through 17 Years Receiving Standard Intravenous Anti-Infective Treatment For Bacterial Infections
Brief Title: Study Of Dalbavancin Drug Levels Achieved In Hospitalized Adolescents Who Are Receiving Antibiotic Therapy For Bacterial Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A8841004
Record Dates: First submitted 2008-05-09; First posted 2008-05-15 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Bacterial Infections
Keywords: dalbavancin adolescent subjects
MeSH Terms: conditions — Bacterial Infections | interventions — dalbavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dalbavancin

INTERVENTIONS:
Drug: Dalbavancin — Subjects weighing > 60 Kg: 1 gram IV single dose Subjects weighing < 60 Kg: 15 mg/Kg IV

SUMMARY:
Adolescent subjects hospitalized for the treatment of bacterial infections will be given 1 gram of dalbavancin through their veins and levels of dalbavancin in blood and urine will be measured at different time points. Safety labs will also be checked on a regular basis to assess the safety of dalbavancin.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 17 year old adolescents hospitalized for the treatment of bacterial infections.

Exclusion Criteria:

* Patients being treated with vancomycin.
* Patients with liver and kidney failure.
* Pregnant female subjects.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Plasma - Cmax, Tmax, AUClast, AUCinf, AUC(48) (as data permit), t1/2 (as data permit), CL, Vss. Urine - Ae48, Ae48% and CLR. | 56 days

SECONDARY OUTCOMES:
Safety assessments: adverse event monitoring; clinical laboratory tests (hematology, serum chemistry, and urinalysis); ECGs; blood pressure and pulse rate determinations; weight and physical examination. | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Cleveland, Ohio

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8841004&StudyName=Study%20Of%20Dalbavancin%20Drug%20Levels%20Achieved%20In%20Hospitalized%20Adolescents%20Who%20Are%20Receiving%20Antibiotic%20Therapy%20For%20Bacterial%20Infections